CLINICAL TRIAL: NCT04801225
Title: Early Feasibility Clinical Study of the Nervive VitalFlow Stimulation System for Treatment of Acute Ischemic Stroke Patients
Brief Title: Early Feasibility Study of the Nervive VitalFlow Stimulation for Acute Ischemic Stroke Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company assets sold. NIH NINDS Grant discontinued.
Sponsor: Nervive, Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV-CP-2020-001; 4U44NS094307 (NIH)
Record Dates: First submitted 2021-03-04; First posted 2021-03-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- VItalFlow Stimulation Treatment (Experimental): Enrolled subjects shall receive a VitalFlow stimulation after other standard-of-care treatments are initiated. VitalFlow treatment is initiated by powering on the System and positioning the two (Left and Right) VItalFlow coils on each side of the head (by the ear).
  The operator controls the VItalFlow Stimulation through the accompanying console with simple button operation. Once treatment is initiated, the VitalFlow provides continuous, biphasic pulses at a preset power cycle with the total treatment time under 5 min (fixed time). After treatment is completed, the coils are removed and replaced on the VitalFlow System.
  Interventions: Device: Non-invasive electromagnetic stimulation for acute stroke treatment

INTERVENTIONS:
Device: Non-invasive electromagnetic stimulation for acute stroke treatment — Bilateral electromagnetic stimulation to improve blood flow in ischemic regions of acute stroke as an adjunct to current standard-of-care
  Other Names: Nervive VitalFlow Stimulator; VitalFlow

SUMMARY:
This Early Feasibility Study (EFS) is a multi-center, open-label single-arm study in 10 acute ischemic stroke (AIS) patients treated with VitalFlow-IS stimulation within 6 hours of symptom onset. The purpose of the EFS is to evaluate initial clinical safety and device functionality in the clinical workflow setting for treatment of acute ischemic stroke patients that will inform design modifications and/or user interface in preparation for next steps consisting of (1) a full safety/feasibility clinical study and (2) randomized controlled pivotal trial with a surrogate endpoint (expedited Premarket Approval (PMA) pathway).

ELIGIBILITY:
Inclusion Criteria:

* Time last known normal within 4.5 hours of presentation for enrollment

  * Allows 1.5 hours for pre-stimulation study procedures to maintain a 6-hour therapeutic window
  * IV rtPA and Endovascular Treatment (EVT) permissible if not inappropriately delayed by study procedures
* Age 18-85 years
* Diagnosis of ischemic stroke in the anterior circulation
* NIHSS at baseline 4-20
* Creatinine < 1.7 mg/dL
* Signed informed consent by patient/Legally Authorized Representative (LAR)

Exclusion Criteria:

* Pre-stroke disability Modified Rankin Score (mRS) between 2-6
* Inability to communicate sufficiently to participate in study procedures
* Neuroimaging with intracranial hemorrhage, severe brain edema, or ASPECTS <5
* Known or newly-discovered aneurysm or arteriovenous malformation (AVM)
* Intracranial mass lesion, infection, or other reason to suspect increased intracranial pressure
* Metallic foreign bodies or implanted devices in the head or neck, including tattoos
* Cardiac, vagal nerve, or intracranial neural stimulation device
* Cochlear implant or implanted hearing aid
* Potential for delay in intravenous rtPA or endovascular therapy due to study procedures

  * Intravenous (IV) rtPA: Stimulation might be delivered during the rtPA infusion period
  * EVT: Stimulation might be performed while EVT team is mobilized
* Seizure concurrent to stroke, or history of seizures, epilepsy, or recurrent syncopal events.
* History of neuropathy (including facial nerve injury), carotid surgery, or vagotomy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Rate of device-related adverse events | 90 days post-procedure
  Rate of device-related adverse events
Feasibility of device use in the Clinical Environment as assessed by User Survey | 1-7 days post-procedure
  To demonstrate feasibility, device must have been able to be setup, deployed, and administer treatment without significant difficulty for each study subject, as recorded by the Investigator on the User Survey.

SECONDARY OUTCOMES:
Exploratory - Rate of change in core volume as measured by Computed Tomography Perfusion | 2-4 hours post-procedure
  Change in core volumes as measured by CTP at pre-stimulation vs 2-4 hours post-stimulation. Being evaluated for potential use as surrogates in future studies.
Exploratory - Rate of change in penumbra volume as measured by Computed Tomography Perfusion | 2-4 hours post-procedure
  Change in penumbra volume as measured by CTP at pre-stimulation vs 2-4 hours post-stimulation. Being evaluated for potential use as surrogates in future studies.
Exploratory - Rate of change in collateral blood flow as measured by Computed Tomography Perfusion | 2-4 hours post-procedure
  Change in collateral blood flow as measured by CTP at pre-stimulation vs 2-4 hours post-stimulation. Being evaluated for potential use as surrogates in future studies.
Exploratory - Rate of change in occlusion status as measured by Computed Tomography Perfusion | 2-4 hours post-procedure
  Change in occlusion status as measured by CTP at pre-stimulation vs 2-4 hours post-stimulation. Being evaluated for potential use as surrogates in future studies.
Exploratory - Difference in baseline core volume on CTP compared to 24 hour MRI final infarct volume | 24 hours post-procedure
  Difference in baseline core volume on CTP compared to 24 hour MRI final infarct volume. Being evaluated for potential use as surrogates in future studies.
Exploratory - Change in National Institute of Health Stroke Scale (NIHSS) - short-term | Pre-procedure, immediately post-procedure, 30, 60, 90, 120, 150, 180, 210, 240 minutes post-procedure
  Change in NIHSS score [range: 1-42, with lower score indicating better outcome] pre to post-stimulation, and every 30 minutes up to 4 hours post-stimulation. Being evaluated for potential use as surrogates in future studies.
Exploratory - Change in National Institute of Health Stroke Scale (NIHSS) - 24 hours | 24 hours post-procedure
  Change in NIHSS score [range: 1-42, with lower score indicating better outcome] pre-stimulation to 24 hours post-stimulation, and every 30 minutes up to 4 hours post-stimulation. Being evaluated for potential use as surrogates in future studies.
Exploratory - Patient Outcome as determined by National Institute of Health Stroke Scale (NIHSS) | 90 days post-procedure
  NIHSS score [range: 1-42, with lower score indicating better outcome] at 90 days post-procedure. Being evaluated for potential use as surrogates in future studies.
Exploratory - Patient Outcome as determined by Modified Rankin Scale (mRS) | 90 days post-procedure
  mRS score [range: 0-6, with lower score indicating better outcome] at 90 days post-procedure. Being evaluated for potential use as surrogates in future studies.
Exploratory - Final change in infarct growth - CTP (CBF<30%) at pre-stimulation vs MRI-DWI lesion at 24 hours | 24 hours post-procedure
  Final change in infarct growth - CTP (CBF<30%) at pre-stimulation vs MRI-DWI lesion at 24 hours. Being evaluated for potential use as surrogates in future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Harrington, MS, Study Director — Nervive, Inc.; Emilio Sacristan, PhD, Study Director — Nervive, Inc.; Ken Uchino, MD, Principal Investigator — The Cleveland Clinic; Jon Schrock, MD, Principal Investigator — MetroHealth System, Ohio
Locations (2):
- United States (2):
  - MetroHealth, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No